CLINICAL TRIAL: NCT05848219
Title: Healthcare Resource Utilization and Costs in Metastatic Melanoma Patients Initiated Dabrafenib + Trametinib and Encorafenib + Binimetinib
Status: Terminated | Type: Observational
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212AUS59
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Dabrafenib + trametinib (dab/tram): Patients with a first diagnosis of metastatic melanoma, who received dab/tram in the United States
- Encorafenib + binimetinib (enco/bini): Patients with a first diagnosis of metastatic melanoma, who received enco/bini in the United States

SUMMARY:
This was a retrospective cohort study using the MarketScan health care administrative claim databases: Truven Health Analytics' MarketScan Commercial Claims and Encounters; MarketScan Medicare Supplement and Coordination of Benefit. We conducted this analysis using the most recent available data from the MarketScan database at the time of analysis, which was 01 June 2018 to 31 December 2020. We initiated this analysis from 01 June 2018 as encorafenib + binimetinib (enco/bini) was approved for patients with unresectable or metastatic melanoma with BRAF mutation at this time.

ELIGIBILITY:
Inclusion Criteria:

* At least one diagnosis of malignant melanoma (The International Classification of Diseases, 9th Revision [ICD-9] codes: 172.0-172.9 or V10.82; ICD-10 codes: C43.0 C43.10 C43.20 C43.30 C43.31 C43.39 C43.4 C43.59 C43.60 C43.70 C43.8 C43.9 D03.0 D03.10 D03.11 D03.12 D03.20 D03.21 D03.22 D03.30 D03.39 D03.4 D03.51 D03.52 D03.59 D03.60 D03.61 D03.62 D03.70 D03.71 D03.72 D03.8 D03.9 Z85.820) in the study period.
* A diagnosis of metastasis (ICD-9 196.x, 197.x, 198.x, 199.x & ICD-10 C77.xx, ICD-10 C78.xx, ICD-10 C79.xx, ICD-10 C80.xx) within 30 days before or 60 days after their malignant melanoma diagnosis.
* A prescription (pharmacy or medical claim) of enco/bini or dab/tram as a 1L therapy after the metastatic melanoma diagnosis date.
* At least ≥18 years as of the index date.
* At least 6 months of continuous enrollment before index date and 6 months after index date.

Exclusion Criteria:

* Patients with a diagnosis of other primary malignancy (ICD-9: 140.xx-165.xx, 170.xx-171.xx, 173.xx-195.xx, 200.xx-208.xx; ICD-10: C00.x - C14.x, C41.x, C49.x, C50, C51) during the 6 months pre-index period.
* Patients with pregnancy (ICD-9: 630.xx-679.xx, V22.xx-V24.xx, V27.xx-V28.xx; ICD-10: O00 - O99) any time during the study period.
* Patients with more than one melanoma-related drug prescription other than the index drug, on the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
All-cause healthcare resource utilization (HCRU) among patients treated with dab/tram versus enco/bini | Up to 2.5 years
All-cause healthcare costs among patients treated with dab/tram versus enco/bini | Up to 2.5 years
Melanoma-specific HCRU among patients treated with dab/tram versus enco/bini | Up to 2.5 years
Melanoma-specific healthcare costs among patients treated with dab/tram versus enco/bini | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, East Hanover, New Jersey, United States